CLINICAL TRIAL: NCT03827538
Title: Endobronchial Valves Positioning Effects On Diaphragm Function In Patients With Lung Hyperinflation - EVELHYN
Brief Title: Endobronchial Valves Positioning Effects On Diaphragm Function In Patients With Lung Hyperinflation
Acronym: EVELHYN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio 2
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Diaphragm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective study aims at evaluating diaphragmatic function before and after endobronchial valves positioning in a COPD patients with lung hyperinflation.

DETAILED DESCRIPTION:
Data obtained from clinical and bimolecular studies have showed that chronic obstructive pulmonary disease (COPD) patients might present higher rates of diaphragm function impairment when compared to age and sex matched healthy controls. The potential mechanisms of injury have been found in regional stresses and strains due to disadvantageous muscle geometry, increased workload during exertion, mechanical stress and metabolic factors (i.e., increased protease activity, free radicals, oxidation). In particular emphysema, with the breakdown of elastic alveolar tissue, leads to increased lung compliance and gas trapping. Lung hyperinflation with amplified dynamic elastance and intrinsic positive end expiratory pressure (PEEPi) limit the diaphragmatic excursion capacity. Moreover both end expiratory lung volume (EELV) and residual volume (RV) increase, shifting tidal breathing (Vt) towards the right side of the pressure-volume curve and imposing higher intra-thoracic pressures to maintain an adequate Vt. Furthermore it has been showed that in COPD patients experiencing frequent exacerbations the maximum pressure produced by diaphragm contraction seems significantly lower as compared to non-COPD subjects, independently on the nature of the tests used for assessment (both volitional - Pdi at Total Lung Capacity (TLC) or Pdi sniff- or non volitional - phrenic nerve stimulation). Thus the reduction of diaphragm maximal performances might be explained by muscle shortening and mechanical impairment following the onset of progressive lung hyperinflation. Lung hyperinflation worsens with exercise leading to breathlessness and is associated with reduced physical activity and reduced survival. Inhaled bronchodilator medications have only modest impacts on symptoms and do not alter the natural history of the disease. In selected patients with a heterogeneous pattern of emphysema, surgical resection can be targeted at the worst affected areas of lung tissue, which contribute disproportionately to gas trapping and hyperinflation, and so improve respiratory mechanics. Lung volume reduction surgery in selected patients (LVRS) improves symptoms and prolongs survival but can be associated with significant morbidity and a risk of death, with a cost per quality adjusted life year (QALY) of at least $40 000.

A more recent approach has been to use endobronchial valves to occlude the airways supplying the worst affected part of the lung. This is intended to cause atelectasis in the target lobe, with a similar impact on the function of the rest of the lung as seen in LVRS. Several trials have demonstrated that endobronchial valve treatment in patients with emphysema can lead to improvements in symptoms, lung function and exercise capacity reductions in dynamic hyperinflation and improvements in oxygen kinetics and chest wall synchrony. While studies on surgical lung volume reduction have demonstrated improvement in diaphragmatic muscle function no studies have investigated the effects of endobronchial valves positioning on diaphragm performance in patients with lung hyperinflation.

Several methods have been used to evaluate diaphragmatic contractile activity. Among these, the standard reference is represented by the measurement of trans-diaphragmatic (Pdi) pressure expressed by the difference between pleural (or esophageal [Pes]) and abdominal (or gastric [Pgas]) pressures through nasogastric probes equipped with pressure sensors. However, such methods are still far from routine clinical practice, thus highlighting the need for simple and accurate methods to assess diaphragmatic performance. In last years the ultrasound (US) evaluation of the diaphragmatic function has been developing in the field of intensive care as a tool to estimate patient's work of breathing during ventilation. In a recently published study on 75 patients with AECOPD requiring mechanical ventilation, we showed a complete correlation between US assessment and Pdi measurements at maximal inspiration in evaluating diaphragm function. In particular we demonstrated that changes of the diaphragm thickness (ΔTdi) < 20% during tidal volume has the same accuracy of transdiaphragmatic pressure in identifying diaphragm impairment. Furthermore we investigated the US evaluation of the diaphragm in patients with amyotrophic lateral sclerosis (ALS) through the ΔTmax index (the ratio between diaphragm thickness at the end of Vt and after maximal inspiration up to total lung capacity). We found that ΔTmax strongly correlates with respiratory functions tests with high accuracy in identifying subjects with FVC <50% of predicted value. Moreover in a recently published study, Bernardi and coworkers presented a non invasive technique to measure PEEPi in COPD patients, through the US assessment of the time latency (msec) between the onset of diaphragm contraction on US and the onset of inspiratory flow (28).

This prospective study aims at evaluating diaphragmatic function before and after endobronchial valves positioning in a COPD patients with lung hyperinflation.

Materials and methods Study population and setting This prospective explorative observational cohort study will be carried out in the Thoracic Endoscopic Unit (TEU) of the University Hospital of Modena Italy over a 24-month period once approval from the local Ethics Committee of Modena will be obtained. Written informed consent to participate to the study will be obtained by all enrolled patients patient.

Patients will be eligible if admitted to the TEU for intervention of endobronchial valves positioning due to documented lung hyperinflation.

Exclusion criteria will include previously documented diaphragmatic dysfunction, the presence of neuromuscular diseases or other forms of myopathy.

All patients will be treated according to the best current clinical practice by the TEU staff, which will be blinded to the purpose of the study.

General measures At enrollment respiratory clinical variables (age, sex, diagnosis and stage, body mass index, smoke habits, comorbidities, previous treatment with systemic steroids) and respiratory function test values will be recorded.

Study procedures A respiratory physician with high expertise in chest US will perform a US assessment of the diaphragm before and after endobronchial valves placement. Motility of the diaphragm is assessed with a B-mode US device (GE Vivid 7, Yorba Linda, CA, USA) connected to a 7-12 MHz linear probe. Measurements are performed in supine position with an average inclination of 45°. The position of the probe is set to obtain the best view of the zone of apposition of the diaphragm, located between the mid-axillary and the posterior axillary line. The diaphragm is identified as a three-layer structure consisting of one relatively non-echogenic muscle layer coated in two echogenic lines determined by peritoneal serosa and diaphragmatic pleura. Diaphragm thickness is measured bilaterally at end-inspiration and end-expiration. The US images will be stored in electronic or paper format by an examiner unaware of the purpose of the study.

In particular the following measurements will be performed:

* ΔTd: change in diaphragm thickness (Tdi) during inspiration starting from FRC to Vt = [(end-inspiratory Tdi - end-expiratory Tdi) / end-expiratory Tdi] X 100)
* ΔTmax: ratio between Tdi at the end of Vt and Tdi after maximal inspiration up to TLC = end-inspiratory Vt Tdi / end-inspiratory TLC Tdi.
* PEEPiecho: P0.1Mx(TLAT,US/100). TLAT = time latency (msec) between the onset of diaphragm contraction on ultrasound and the onset of inspiratory flow; P0.1M = mouth occlusion pressure at 100ms, an estimate of the effort a patient must make to generate the inspiratory flow. It is measured using a unidirectional valve, occluded during expiration so that the P0.1M is measured from functional residual capacity (FRC).
* US measurement of maximal diaphragmatic inspiratory excursion measured in right subcostal window.

An assessment of maximal expiratory pressure (MEP) and maximal inspiratory pressure (MIP), and sniff inspiratory nasal pressure (SNIP), will be performed before and after endobronchial valves placement by a respiratory function technician unaware of the purpose of the study.

Each outcome measurements will be performed 24 hours, 48 hours, 7 days, 30 days, 60 days and 90 days after endobronchial valves placement.

Statistical analysis The statistical package GraphPad Prism 7.0 (GraphPad Software, Inc. La Jolla, CA, USA) will be used for analysis. Descriptive statistics for continuous variables will be presented as mean values ± standard deviation (SD) or associated to interquartile range. The nonparametric Wilcoxon test (Mann-Whitney) and t student test will be used for comparison of continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* patient admission for intervention for endobronchial valves positioning due to documented lung hyperinflation.

Exclusion Criteria:

* previously documented diaphragmatic dysfunction
* the presence of neuromuscular diseases or other forms of myopathy
* pregnancy
* lack of collaboration in performing functional diaphragmatic tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diaphrgam function test modification after ELVR | 90 days
  Ultrasound assessed ΔTdi values change after ELVR
Diaphrgam fatigue test modification after ELVR | 90 days
  Ultrasound assessed ΔTmax values change after ELVR
Diaphrgam performance test modification after ELVR | 90 days
  Ultrasound assessed PEEPiecho values change after ELVR
Diaphrgam motion test modification after ELVR | 90 days
  US assessed maximal diaphragmatic inspiratory excursion after ELVR

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Modena Policlinico, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided